CLINICAL TRIAL: NCT05810480
Title: Prospective Multicenter Study: PredIcting SterOid DepeNdEnt LivEr Injury (PIONEER) with Polyreactive Immunoglobulin G
Brief Title: PredIcting SterOid DepeNdEnt LivEr InjuRy with Polyreactive Immunoglobulin G
Acronym: PIONEER
Status: Recruiting | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Engel, Bastian Dr., Principal Investigator, Hannover Medical School
Other Study IDs: PIONEER
Record Dates: First submitted 2023-03-28; First posted 2023-04-12 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Autoimmune Hepatitis; Autoimmune Liver Disease
MeSH Terms: conditions — Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Autoimmune Hepatitis: This group includes patients with a diagnosis of Autoimmune Hepatitis according to the simplified diagnostic criteria by Hennes et al. made by the local treating physician. The diagnosis of autoimmune hepatitis additionally requires steroid dependency > six months for this study to discriminate Autoimmune Hepatitis from autoimmune like drug-induced liver injury (DILI) which are hard to discriminate at diagnosis and with the latter often being treating with a short course of corticosteroids less than six months. One serum sample will be stored for anonymized evaluation of serum autoantibodies
  Interventions: Diagnostic Test: polyreactive immunoglobulin G
- non-autoimmune hepatitis liver disease: This group includes patients with a diagnosis of any non-viral liver disease that is not autoimmune hepatitis and whose diagnosis necessitated a diagnostic liver biopsy in the work-up of the liver disease for local care. One serum sample will be stored for anonymized evaluation of serum autoantibodies
  Interventions: Diagnostic Test: polyreactive immunoglobulin G

INTERVENTIONS:
Diagnostic Test: polyreactive immunoglobulin G — Polyreactive immunoglobulin G will be tested centralized in Hannover as published (Taubert, Engel et al., Hepatology, 2022). The current standard diagnostic autoantibodies (e.g. ANA, anti-SMA, anti-LKM, anti-LC1, anti-SLA/L) will be tested centrally in Hannover according to current guidelines.
  Other Names: Conventional diagnostic autoantibodies

SUMMARY:
The investigators identified polyreactive immunoglobulin G (pIgG) in adults (published in Hepatology: https://doi.org/10.1002/hep.32134) and children (in preparation). Quantification of these pIgG using a "home-made" ELISA facilitates the diagnosis of autoimmune hepatitis (AIH) as compared to non-AIH liver diseases and healthy controls. Positivity for pIgG was independent from ANA/SMA positivity and equally diagnostic for AIH even when conventional autoantibodies (ANA/SMA/SLA/LKM) were negative.

Additionally, the frequency of pIgG was lower than conventional autoantibodies (ANA, SMA) in vaccinia/drug associated severe liver injury in a retrospective multicenter study after Covid-19 vaccination (https://doi.org/10.1016/j.jhepr.2022.100605).

Aims of the study The study aims to evaluate the diagnostic capacity of pIgG to predict AIH in comparison to other liver diseases prospectively. To avoid diagnostic inaccuracy between AIH with long-term need for an immunosuppression and drug induced liver injury with autoimmune features, which can be indistinguishable from AIH at baseline and which has a very low relapse rate after a short steroid course, a follow-up after six months is obligatory for inclusion.

Therefore, the investigators will collect one serum sample from every patient (without immunosuppressive treatment) that presents to the respective hospital for evaluation of liver disease by liver biopsy within one year after initiation of the study and that provided written informed consent. Follow-up for evaluation of steroid dependency at six months after diagnosis is obligatory.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic liver biopsy for the work-up of any liver disease
* Informed consent
* Definition of any liver disease according to current societal guidelines

Exclusion Criteria:

* No ongoing immunosuppression at the liver biopsy or prior to the liver biopsy
* Liver biopsies for the grading or staging of an already known liver disease (e.g. non-alcoholic fatty liver disease (NAFLD), Hepatitis B/D Virus Infections (HBV/HDV Infection), …)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient that presents to the respective hospital for evaluation of a so far unknown-liver disease and consents is eligible if the treating physician orders a liver biopsy for the diagnostic evaluation of the liver disease. Patients are not eligible if a liver biopsy is performed for staging or grading of an already known liver disease or if the patient is treated with immunosuppressive drugs at the time of the liver biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Prediction of steroid dependent hepatitis | Assessment of steroid dependency at six months after enrollment
  Prediction of steroid dependent hepatitis by elevated polyreactive immunoglobulin G

SECONDARY OUTCOMES:
Diagnostic discrimination between AIH and DILI by polyreactive IgG | At enrollment
Prediction of steroid dependent hepatitis by any other autoantibody | Assessment of steroid dependency at six months after enrollment
  Prediction of steroid dependent hepatitis by any other elevated conventional autoantibody according to current guidelines (European Association for the study of the liver: EASL, American Association for the Study of Liver Diseases: AASLD)

OTHER OUTCOMES:
Concordance of different testing methods for autoantibodies | At enrollment
  Different methodology to assess presence of autoantibodies (e.g. ELISA, Immunofluorescence on tissue sections) will be tested head-to-head for their diagnostic capacity

CONTACTS AND LOCATIONS:
Overall Officials: Bastian Engel, Dr., Principal Investigator — Hannover Medical School; Richard Taubert, Dr., Principal Investigator — Hannover Medical School
Locations (8):
- Germany (8):
  - University Medical Centre Aachen, Aachen
  - University Hospital Bonn, Bonn
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Hannover Medical School, Hanover
  - University Medical Center Heidelberg, Heidelberg
  - University Hospital Schleswig-Holstein, Location Lübeck, Lübeck
  - University Hospital Magdeburg, Magdeburg
  - Rostock University Medical Centre, Rostock

IPD SHARING:
Plan to Share IPD: No
IPD are not shared with collaborators. Data, in general, is only provided anonymized by contributing centers.

REFERENCES:
- [Background] Taubert R, Engel B, Diestelhorst J, Hupa-Breier KL, Behrendt P, Baerlecken NT, Suhs KW, Janik MK, Zachou K, Sebode M, Schramm C, Londono MC, Habes S; UK-AIH Consortium; Oo YH, Lalanne C, Pape S, Schubert M, Hust M, Dubel S, Thevis M, Jonigk D, Beimdiek J, Buettner FFR, Drenth JPH, Muratori L, Adams DH, Dyson JK, Renand A, Graupera I, Lohse AW, Dalekos GN, Milkiewicz P, Stangel M, Maasoumy B, Witte T, Wedemeyer H, Manns MP, Jaeckel E. Quantification of polyreactive immunoglobulin G facilitates the diagnosis of autoimmune hepatitis. Hepatology. 2022 Jan;75(1):13-27. doi: 10.1002/hep.32134. Epub 2021 Dec 5. PMID 34473365